CLINICAL TRIAL: NCT06928337
Title: CHLOE Oocyte Data Collection Protocol
Brief Title: Data Collection Protocol for the Development of CHLOE-OQ, an AI Model for Assessing Oocytes Quality.
Status: Recruiting | Type: Observational
Sponsor: Fairtility (Industry)
Responsible Party: Sponsor
Other Study IDs: FRT-24-14
Record Dates: First submitted 2025-03-27; First posted 2025-04-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: AI evaluation of oocytes. — AI evaluation of oocytes inside a time-lapse incubator.

SUMMARY:
This data collection protocol is aimed to allow the reliable and robust development (training, verification, and validations) of CHLOE technology-based applications as well as improve the machine learning stage of released devices/applications. Additionally, a simulated use assessments will be conducted to ensure the correct and easy use of the CHLOE applications.

DETAILED DESCRIPTION:
The CHLOE-OQ Data Collection Protocol is designed to support the reliable and robust development of the CHLOE technology-based application, ensuring their accuracy and effectiveness in assessing oocyte quality. This protocol facilitates the entire AI model development lifecycle, including training, verification, and validation, to enhance the performance and reliability of machine learning algorithms integrated into the CHLOE application.

Additionally, the protocol aims to refine the machine learning stage of the already released OQ applications by incorporating new data and improving model performance over time. A key component of this process includes simulated use assessments, which are conducted to evaluate the usability, accuracy, and overall functionality of CHLOE applications in real-world clinical settings by means of a questionnaire for embryologist using CHLOE. These assessments ensure that the technology is not only scientifically sound but also user-friendly, making it easier for embryologists to integrate CHLOE applications into their workflow efficiently.

By adhering to this structured data collection protocol, the CHLOE application can continuously evolve, maintaining high standards of performance and usability in the assessment of oocyte quality.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years of age.
* Embryos or eggs cultured in a time-lapse incubator connected to CHLOE Embryo Viewer.

Exclusion Criteria:

* Women with autologous eggs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oocyte donors
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) will be quantified using logistic regression to assess CHLOE OQ's prediction of blastulation. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Wiemer, 704 9079714, Study Chair — klaus.wiemer@fairtility.com
Locations (1):
- The World Egg and Sperm Bank, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided